CLINICAL TRIAL: NCT06851026
Title: Investigating the Effects of Pilates on Body Composition, Posture, and Psychosocial Parameters in Women with and Without Obesity: a Randomized Controlled Study
Brief Title: Pilates Effect on Women with and Without Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sema Arslan Kabasakal, Asisst. Prof., University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023/161; 1919B012224567 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Obesity Prevention; Obesity and Overweight; Exercise; Pilates Exercise
Keywords: exercise; obesity; health; physical fitness; psychology
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: This study follows a randomized, parallel assignment interventional model with an open-label design. Participants were randomly assigned into four groups based on their obesity status and Pilates intervention:
  Pilates group with obesity Pilates group without obesity Control group with obesity Control group without obesity The intervention consisted of an 8-week Pilates program administered to the experimental groups, while control groups did not receive any intervention. The study aimed to examine the effects of Pilates on BMI, fat percentage, posture, emotional eating, social physical anxiety, and self-esteem.
  A mixed-design ANOVA was conducted to analyze the interaction between time (pre-test vs. post-test) and group differences. ANCOVA was used to adjust for baseline differences. Additional analyses, including independent samples t-tests and Chi-Square tests, were performed to assess BMI category changes. The study was conducted with an α-level of 0.05 for statistical significance
Who Masked: Participant, Investigator
Masking Description: The researcher who performed the exercises was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pilates Group with Obesity (Experimental): The obese intervention group received Pilates exercises for 8 weeks.
  Interventions: Other: Pilates Exercise
- Pilates Group without Obesity (Experimental): The non-obese intervention group received Pilates exercises for 8 weeks.
  Interventions: Other: Pilates Exercise
- Control Group with Obesity (No Intervention): The obese control group received no intervention for 8 weeks.
- Control Group without Obesity (No Intervention): The non-obese control group received no intervention for 8 weeks.

INTERVENTIONS:
Other: Pilates Exercise — Pilates exercises were applied for 8 weeks
  Arms: Pilates Group with Obesity; Pilates Group without Obesity

SUMMARY:
Obesity, a health problem, is caused by insufficient physical activity and unhealthy nutrition. For individuals with obesity, non-weight-bearing and enjoyable exercises, such as Pilates, should be implemented as physical activity due to potential pain. This study aims to examine the effects of an 8-week Pilates exercise program on body composition, posture, and psychosocial parameters in individuals with and without obesity. Methods: The study included 58 female participants: 30 individuals with obesity (nPilates = 15; nControl = 15) and 28 individuals without obesity (nPilates = 14; nControl = 14). Participants performed Pilates exercises twice a week for 8 weeks. Body Mass Index (BMI), body fat percentage (BFP), and posture scores were calculated, and from a psychosocial perspective Emotional Eating Scale (EE), Social Physique Anxiety Inventory (SPA), and Self-Esteem Scales (SE) were administered before and after the eight weeks.

DETAILED DESCRIPTION:
There are no studies in the literature examining the effects of Pilates exercises on emotional eating and posture. Additionally, there are no studies examining the effects of Pilates on posture in individuals with obesity. Most studies in the literature have focused on sedentary women; however, no study has specifically examined the effects of Pilates-based exercises on individuals with and without obesity. This study aims to investigate the effects of an 8-week Pilates intervention on postural alignment, BMI, fat percentage, and psychosocial parameters (emotional eating, social physical anxiety, and self-esteem) in individuals with and without obesity. Thus, this study will provide valuable insights into the role of Pilates in weight management, posture correction, and psychosocial well-being among individuals with and without obesity. The study included 58 female participants: 30 individuals with obesity (nPilates = 15; nControl = 15) and 28 individuals without obesity (nPilates = 14; nControl = 14). Participants performed Pilates exercises twice a week for 8 weeks. Body Mass Index (BMI), body fat percentage (BFP), and posture scores were calculated, and from a psychosocial perspective Emotional Eating Scale (EE), Social Physique Anxiety Inventory (SPA), and Self-Esteem Scales (SE) were administered before and after the eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being a sedentary individual and not not doing regular physical activity
* Being 20 years old or older
* Having a BMI of 30 kg/m² or above for inclusion in the group of women with obesity.
* Having a BMI below 30 kg/m² for inclusion in the group of women without obesity.
* Not having any health problems that would prevent participation in exercise.
* Not having undergone surgery affecting the musculoskeletal system within the last year.

Exclusion Criteria:

* Voluntary withdrawal from the study.
* Failure to comply with the required procedures of the study.
* Arbitrary disruption of the exercise schedule more than twice.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 58 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and at the end of 8 weeks
  Difference in BMI before and after the 8-week Pilates intervention. BMI is calculated as weight (kg) divided by height (m²).
Change in Body Fat Percentage | Baseline and at the end of 8 weeks
  Difference in body fat percentage before and after the intervention, assessed using bioelectrical impedance analysis (BIA)
Change in Posture Score | Baseline and at the end of 8 weeks
  Assessed using the New York Posture Rating Scale to evaluate improvements in postural alignment. This assessment is conducted by scoring potential postural changes in 13 different parts of the body. If the person's each parts of body posture is correct, a score of 5 is given; if moderately impaired, a score of 3; and if severely impaired, a score of 1. The total score ranges from a maximum of 65 to a minimum of 13. A higher score indicates better posture alignment.

SECONDARY OUTCOMES:
Changes in Emotional Eating | Baseline and at the end of 8 weeks
  Participants' emotional eating changes were measured with the Emotional Eating Scale. The scale consists of 10 items and is structured in a 4-point Likert format (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always). The scale is scored between 0 and 30. A score of "30" indicates the highest level of emotional eating behavior, while a score of "0" indicates the absence of emotional eating behavior.
Change in Social Physique Anxiety | Baseline and at the end of 8 weeks
  Changes in participants' social physics anxiety levels were measured with The Social Physique Anxiety Inventory. The items in the inventory are answered using a five-point scale (completely false, mostly false, sometimes false, sometimes true, mostly true, completely true). The minimum possible score from the inventory is 12, and the maximum is 60. Higher scores indicate higher levels of anxiety about physical appearance
Change in Self-Esteem | Baseline and at the end of 8 weeks
  The Rosenberg Self-Esteem Scale was used to measure self-esteem. The scale consists of 31 items. The minimum score is 31 and the maximum score is 155. An increase in the score obtained from the scale indicates an increase in self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Arslan Kabasakal, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We attach importance to protecting the confidentiality of data.

REFERENCES:
- [Background] Arslan Kabasakal S, Delice B. Investigating the Effects of Pilates on Body Composition, Posture, and Psychosocial Parameters in Women With and Without Obesity: A Randomized Controlled Study. J Phys Act Health. 2025 Aug 23;22(12):1557-1567. doi: 10.1123/jpah.2024-0498. Print 2025 Dec 1. PMID 40849103
- See also: The dataset supporting the findings of this study is restricted due to privacy concerns. Researchers may request access by contacting [institution/contact details]. — https://sporbilimleri.yalova.edu.tr/